CLINICAL TRIAL: NCT01596361
Title: Verification of a Pharmacogenetic Approach to Customizing Chemotherapy to Asians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/01711
Record Dates: First submitted 2012-04-02; First posted 2012-05-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Interethnic variability in chemotherapy response is becoming increasingly evident, making approaches for customizing chemotherapy treatment to different ethnic populations desirable. At the same time, significant genetic variation has also been observed between ethnic groups, including many germline and somatic pharmacogenetic variants involved in chemotherapy pharmacology. Recently, based on meta-analyses of studies on germline pharmacogenetic variant frequencies and clinical trials, the investigators found that chemotherapy outcomes between Asians and Caucasians colorectal cancer (CRC) patients could potentially be inferred from the frequencies of variants between the ethnic groups and their respective biological functions. In this study, the investigators seek to further clarify the validity of using pharmacogenetic variants to customize chemotherapy between ethnicities through the following specific aims: (1) To verify the differences observed in the frequency of germline pharmacogenetic variants related to chemotherapy between Asian and Caucasian CRC patients, (2) To test whether variations in the frequency of somatic pharmacogenetic gene mutations between Asian and Caucasian CRC patients could be used to infer differences in clinical outcomes between the two ethnicities. (3) (4) For Aim 1, DNA samples from approximately 1000 Asian and Caucasian CRC patients each will be analyzed for the frequency of a panel of germline pharmacogenetic variants identified in our meta-analyses using high-throughput methodology. For Aim 2, meta-analyses will be performed on pharmacogenetic studies and clinical trials to establish the relative frequencies of somatic variants and clinical outcomes in Asian and Caucasian CRC patients. These frequencies will be verified on the same series of DNA samples used in Aim 1. The clinical outcomes inferred from the frequency differences and biological functions will then be compared to those summarized from clinical trials. This data could provide a basis for developing a rational approach to customizing chemotherapy in non-Caucasian populations and improve assessment of drug feasibility in different ethnic populations.If validated, this working hypothesis would be of high clinical interest, giving the opportunity to use this as a DNA prognosis biomarker in CRC.

Pharmacogenetic frequencies could be a potentially useful approach for predicting likely chemotherapy outcomes in non-Caucasian populations

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples will be obtained from the Tissue Repository, National University Hospital, St. John of God Hospital, Perth, Australia and Kanazawa University, Japan.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Verify the differences observed in the frequency of germline pharmacogenetic variants related to chemotherapy between Asian and Caucasian CRC patients

SECONDARY OUTCOMES:
Testing the variations in the frequency of somatic pharmacogenetic gene mutations between Asian and Caucasian CRC patients could be used to infer differences in clinical outcomes between the two ethnicities.
Characterise the deletion status of heat shock protein molecules and determine the association between heat shock protein deletion status and clinico-pathological outcomes in Asian and Caucasian patients with CRC

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore